CLINICAL TRIAL: NCT03352037
Title: 18F-FDG PET/MR Imaging for Differentiation of Serous From Non-Serous Pancreatic Cystic Neoplasms: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN-16-6058
Record Dates: First submitted 2017-11-13; First posted 2017-11-24 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Cystic Neoplasms
MeSH Terms: interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): In this project, there is only one study group which comprises of patients with pancreatic cystic neoplasms who will undergo pancreatic PET/MRI.
  Interventions: Diagnostic Test: PET scan

INTERVENTIONS:
Diagnostic Test: PET scan — Patients with known pancreatic cystic lesions requiring MR imaging for lesion characterization for clinical evaluation will be recruited to undergo 18F-FDG PET/MR imaging after written informed consent.

SUMMARY:
The overlap of morphological imaging features results in many incidentally detected pancreatic cystic neoplasms going undiagnosed, including benign serous cystic neoplasms (SCN) and potentially malignant mucinous lesions (nonserous). The diagnostic ambiguity then lead to invasive procedures such as endoscopic ultrasonography (EUS), unwarranted surgical resection on SCN lesions or the need for long term periodic surveillance with delayed diagnosis of potentially malignant nonserous lesions. Therefore, precise differentiation of SCN from nonserous cystic neoplasms is highly desirable.

The 18F-fluorodeoxyglucose (FDG) accumulation in tumor cells, which is induced by high expression of glucose transporter proteins (mainly include GLUT-1 and -3), can be used to discriminate malignant and benign pancreatic cystic tumors in positron emission tomography (PET) imaging. GLUT-1 expression has also been documented in benign SCN while no such evidence exists in potentially malignant nonserous cystic neoplasms. Based on this evidence, investigators will conduct a pilot study to evaluate if integrated 18F-FDG PET/MR imaging with simultaneous MR and PET acquisition is helpful in differentiation of SCN from nonserous lesions.

ELIGIBILITY:
Inclusion Criteria:

-Patients with known pancreatic cystic lesions, including suspected pancreatic serous cystic neoplasms and non-serous cystic neoplasms

Exclusion criteria:

* General Contraindications to MRI such as pacemaker, brain aneurysm clip etc. -
* Pregnancy
* Age below 18 years
* Estimated GFR (eGFR < 30 mL/min)
* MRI contrast allergy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Investigation of 18F-FDG PET/MRI efficacy in differentiating pancreatic cystic neoplasms | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Jhaveri, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada